CLINICAL TRIAL: NCT01573273
Title: Oxytocin in Cocaine Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Associate Professor of Psychiatry, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 00016890
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Cocaine Dependence
Keywords: cocaine; substance abuse; drug abuse; cocaine dependence; drug addiction
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- TSST Women Oxytocin (Experimental): Cocaine-dependent women received 40 IUs of intranasal oxytocin prior to completing a Social Stress Task.
  Interventions: Drug: Oxytocin
- TSST Women Placebo (Placebo Comparator): Cocaine-dependent women received intranasal saline prior to completing a Social Stress Task.
  Interventions: Drug: Saline
- MRI 1 Women Oxytocin (Experimental): Cocaine-dependent women received 40 IUs of intranasal oxytocin prior to completing the first of two fMRI cue-exposure tasks.
  Interventions: Drug: Oxytocin
- MRI 1 Women Placebo (Placebo Comparator): Cocaine-dependent women received intranasal saline prior to completing the first of two fMRI cue-exposure tasks.
  Interventions: Drug: Saline
- MRI 2 Women Oxytocin (Experimental): Cocaine-dependent women received 40 IUs of intranasal oxytocin prior to completing the second of two fMRI cue-exposure tasks.
  Interventions: Drug: Oxytocin
- MRI 2 Women Placebo (Placebo Comparator): Cocaine-dependent women received intranasal saline prior to completing the second of two fMRI cue-exposure tasks.
  Interventions: Drug: Saline
- TSST Men Oxytocin (Experimental): Cocaine-dependent men received 40 IUs of intranasal oxytocin prior to completing a Social Stress Task.
  Interventions: Drug: Oxytocin
- TSST Men Placebo (Placebo Comparator): Cocaine-dependent men received intranasal saline prior to completing a Social Stress Task.
  Interventions: Drug: Saline
- MRI I Men Oxytocin (Experimental): Cocaine-dependent men received 40 IUs of intranasal oxytocin prior to completing the first of two fMRI cue-exposure tasks.
  Interventions: Drug: Oxytocin
- MRI I Men Placebo (Placebo Comparator): Cocaine-dependent men received intranasal saline prior to completing the first of two fMRI cue-exposure tasks.
  Interventions: Drug: Saline
- MRI 2 Men Oxytocin (Experimental): Cocaine-dependent men received 40 IUs of intranasal oxytocin prior to completing the second of two fMRI cue-exposure tasks.
  Interventions: Drug: Oxytocin
- MRI 2 Men Placebo (Placebo Comparator): Cocaine-dependent men received intranasal saline prior to completing the second of two fMRI cue-exposure tasks.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Oxytocin — intranasal administration, 40 IUs
  Other Names: pitocin
  Arms: MRI 1 Women Oxytocin; MRI 2 Men Oxytocin; MRI 2 Women Oxytocin; MRI I Men Oxytocin; TSST Men Oxytocin; TSST Women Oxytocin
Drug: Saline — intranasal administration, 40 IUs
  Other Names: pitocin
  Arms: MRI 1 Women Placebo; MRI 2 Men Placebo; MRI 2 Women Placebo; MRI I Men Placebo; TSST Men Placebo; TSST Women Placebo

SUMMARY:
Stress is likely involved in relapse to cocaine use. This project will investigate the role oxytocin may play in the stress response in cocaine-dependent men and women and examine how oxytocin may impact brain activity in individuals exposed to cocaine-related cues.

DETAILED DESCRIPTION:
Stress is an important predictor of relapse, and targeting stress-activated pathways may lead to therapeutic advancements in the treatment of substance use disorders. Oxytocin has been shown to promote trust, social bonding, and calmness; however, its potential effects have not been explored in cocaine-dependent individuals. Oxytocin receptors have been localized to brain regions that are activated by drug-paired cues and preclinical studies have shown that oxytocin attenuates the acute and long-term behavioral effects of psychostimulants. However, little is known about the role of oxytocin in mediating the affective response to cocaine-paired cues and associated neural activity in cocaine-dependent men and women. This project is a direct evolution from our previous SCOR-supported research. Our work has progressed from characterizing sex/gender differences in response to social stressors and cocaine cues in cocaine-dependent men and women, to our on-going work evaluating whether stress potentiates cue-induced craving and the impact of hormones on this response. The proposed study will investigate the role of oxytocin in the sex/gender differences in stress response and craving in cocaine-dependent individuals and preliminarily explore its therapeutic potential.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Subjects must meet DSM-IV criteria for current cocaine dependence (within the past three months). While individuals may also meet criteria for abuse of other substances, they must not meet criteria for dependence on any other substance (except nicotine) within the last 60 days. Alcohol has been known to affect HPA function (Adinoff et al., 1991), however to enhance recruitment efforts individuals with alcohol dependence or abuse will be included in the study if they do not require medically supervised detoxification. Also, due to the high comorbidity of cocaine and marijuana dependence, and limited evidence that marijuana use affects HPA function, subjects with marijuana dependence will be included.
3. Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) for a three-day period immediately prior to the throughout study procedures.
4. Subjects must consent to random assignment.
5. Subjects must consent to participating in study procedures at the ASD and completion of two fMRI scans.

Exclusion Criteria

1. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control (not including hormonal contraceptives).
2. Women who are currently taking, or have taken in the past month, oral or other types of hormonal contraceptives or hormone replacement therapies.
3. Women with premenstrual dysphoric disorder who are outside of the follicular phase.
4. Women who have had a complete hysterectomy or are over 50 over one year post-menopausal, as ovarian hormones will be measured in the study.
5. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect physiological/subjective responses. Neurological exclusions include history of stroke, seizure disorders, multiple sclerosis, Parkinson's disease, and Alzheimer's disease.
6. Subjects with Addison's disease, Cushing's disease or other diseases of the adrenal cortex likely to affect hormonal/neuroendocrine status.
7. Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with subjective measurements.
8. Subjects with current major depressive disorder or post-traumatic stress disorder as these disorders are associated with characteristic changes in stress response.
9. Subjects receiving synthetic glucocorticoid therapy, any exogenous steroid therapy, or treatment with other agents that interfere with hormonal measurements within one month of test session.
10. Subjects taking any mood stabilizers, antipsychotics, benzodiazepines, opiates or opiate antagonists because these may affect test response. Subjects taking SSRI's will be included.
11. Subjects with any acute illness or fever. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
12. Subjects whose height to weight ratio would preclude them from fitting comfortably in the MRI scanner.
13. Subjects who are unwilling or unable to maintain abstinence from alcohol and other drugs of abuse (except nicotine) for three days prior to the stress task procedure.
14. Persons with ferrous metal implants or pacemaker since fMRI will be used.
15. Subjects who are claustrophobic.
16. Subjects with significant psychiatric or medical problems that would impair participation or limit ability to participate in scan.
17. Subjects who require maintenance or acute treatment with any psychoactive medication including anti-seizure medications which could potentially interfere with fMRI.
18. Subjects meeting DSM-IV criteria for substance dependence (other than nicotine, cocaine, alcohol or marijuana) within the past 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-10; Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee McRae-Clark, Pharm.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 112 is the total number of participants randomized. 112 completed the TSST, which was between groups. MRIs were within subjects; 99 completed at least MRI 1. 96 completed MRI's 1 and 2. Data is reported per testing condition.
Period: TSST : Trier Social Stress Task
Arm/Group | TSST Women Oxytocin | TSST Women Placebo | MRI 1 Women Oxytocin | MRI 1 Women Placebo | MRI 2 Women Oxytocin | MRI 2 Women Placebo | TSST Men Oxytocin | TSST Men Placebo | MRI I Men Oxytocin | MRI I Men Placebo | MRI 2 Men Oxytocin | MRI 2 Men Placebo
Started | 24 | 25 | 0 | 0 | 0 | 0 | 32 | 31 | 0 | 0 | 0 | 0
Completed | 24 | 25 | 0 | 0 | 0 | 0 | 32 | 31 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MRI 1
Arm/Group | TSST Women Oxytocin | TSST Women Placebo | MRI 1 Women Oxytocin | MRI 1 Women Placebo | MRI 2 Women Oxytocin | MRI 2 Women Placebo | TSST Men Oxytocin | TSST Men Placebo | MRI I Men Oxytocin | MRI I Men Placebo | MRI 2 Men Oxytocin | MRI 2 Men Placebo
Started | 0 | 0 | 19 | 23 | 0 | 0 | 0 | 0 | 28 | 29 | 0 | 0
Completed | 0 | 0 | 19 | 23 | 0 | 0 | 0 | 0 | 28 | 29 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MRI 2
Arm/Group | TSST Women Oxytocin | TSST Women Placebo | MRI 1 Women Oxytocin | MRI 1 Women Placebo | MRI 2 Women Oxytocin | MRI 2 Women Placebo | TSST Men Oxytocin | TSST Men Placebo | MRI I Men Oxytocin | MRI I Men Placebo | MRI 2 Men Oxytocin | MRI 2 Men Placebo
Started | 0 | 0 | 0 | 0 | 23 | 18 | 0 | 0 | 0 | 0 | 27 | 28
Completed | 0 | 0 | 0 | 0 | 23 | 18 | 0 | 0 | 0 | 0 | 27 | 28
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 112 is the total number of participants randomized to receive Oxytocin or Placebo prior to the TSST.
Groups:
- Cocaine- Dependent Women Oxytocin: Cocaine-dependent women received 40 IUs of intranasal oxytocin prior to completing a Social Stress Task on Day 1, and MRI on Day 2 and an MRI on Day 3. The TSST task was between subjects; the MRI tasks were within subjects.
- Cocaine- Dependent Men Oxytocin: Cocaine-dependent men received 40 IUs of intranasal oxytocin prior to completing a Social Stress Task on Day 1, and MRI on Day 2 and an MRI on Day 3. The TSST task was between subjects; the MRI tasks were within subjects.
- Cocaine- Dependent Women Placebo: Cocaine-dependent women received Placebo prior to completing a Social Stress Task on Day 1, and MRI on Day 2 and an MRI on Day 3. The TSST task was between subjects; the MRI tasks were within subjects.
- Cocaine -Dependent Men Placebo: Cocaine-dependent men received Placebo prior to completing a Social Stress Task on Day 1, an MRI on Day 2 and an MRI on Day 3. The TSST task was between subjects; the MRI tasks were within subjects.
- Total: Total of all reporting groups
Arm/Group | Cocaine- Dependent Women Oxytocin | Cocaine- Dependent Men Oxytocin | Cocaine- Dependent Women Placebo | Cocaine -Dependent Men Placebo | Total
Number analyzed (Participants) | 24 | 32 | 25 | 31 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 32 | 25 | 31 | 112
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 0 | 25 | 0 | 49
  Male | 0 | 32 | 0 | 31 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 18 | 24 | 13 | 24 | 79
  White | 6 | 8 | 11 | 7 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 32 | 25 | 31 | 112

OUTCOME MEASURES:

1. Primary Outcome: Subjective Stress Response TSST
Description: Subjects rated stress levels on a 0-10 Likert Scale where 0 is Not at All and 10 is Extremely so that lower scores indicate lower stress levels.
Time Frame: Subjects rated stress immediately following a Social Stress task on Day 1 of 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TSST Women Oxytocin | TSST Women Placebo | TSST Men Oxytocin | TSST Men Placebo
Number analyzed (Participants) | 24 | 25 | 32 | 31
units on a scale | 5.33 (3.81) | 5.28 (4.09) | 2.05 (2.34) | 2.13 (2.87)

2. Primary Outcome: Subjective Stress Response MRI 1
Description: as for outcome 1
Time Frame: Subjects rated Stress immediately following the first of two MRI scans on Day 2 of 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- MRI 1 Women Oxytocin: Cocaine-dependent women received 40 IUs of intranasal oxytocin prior to completing the first of two MRI scans.
  Oxytocin: intranasal administration, 40 IUs
- MRI 1 Women Placebo: Cocaine-dependent women received intranasal saline prior to completing the first of two MRI scans.
  Saline: intranasal administration, 40 IUs
- MRI 1 Men Oxytocin: Cocaine-dependent men received 40 IUs of intranasal oxytocin prior to completing the first of two MRI scans.
  Oxytocin: intranasal administration, 40 IUs
- MRI 1 Men Placebo: Cocaine-dependent men received intranasal saline prior to completing the first of two MRI scans.
  Saline: intranasal administration, 40 IUs
Arm/Group | MRI 1 Women Oxytocin | MRI 1 Women Placebo | MRI 1 Men Oxytocin | MRI 1 Men Placebo
Number analyzed (Participants) | 19 | 23 | 28 | 29
units on a scale | 2.05 (2.34) | 2.13 (2.87) | 1.75 (2.40) | 2.66 (2.84)

3. Primary Outcome: Subjective Stress Response MRI 2
Description: as for outcome 1
Time Frame: Subjects rated stress immediately following the second of two MRI scans on Day 3 of 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- MRI 2 Women Oxytocin: Cocaine-dependent women received 40 IUs of intranasal oxytocin prior to completing the second of two MRI scans.
  Oxytocin: intranasal administration, 40 IUs
- MRI 2 Women Placebo: Cocaine-dependent women received intranasal saline prior to completing the second of two MRI scans.
  Saline: intranasal administration, 40 IUs
- MRI 2 Men Oxytocin: Cocaine-dependent men received 40 IUs of intranasal oxytocin prior to completing the second of two MRI scans.
  Oxytocin: intranasal administration, 40 IUs
- MRI 2 Men Placebo: Cocaine-dependent men received intranasal saline prior to completing the second of two MRI scans.
  Saline: intranasal administration, 40 IUs
Arm/Group | MRI 2 Women Oxytocin | MRI 2 Women Placebo | MRI 2 Men Oxytocin | MRI 2 Men Placebo
Number analyzed (Participants) | 23 | 18 | 27 | 28
units on a scale | 0.83 (1.67) | 1.83 (2.81) | 1.07 (2.07) | 1.39 (2.06)

4. Secondary Outcome: Subject Cocaine Craving TSST
Description: Subjects rated craving on a 0-10 Likert Scale where 0 is Not at All and 10 is Extremely so that lower scores indicate lower craving.
Time Frame: Subjects rated craving immediately following a Social Stress task on Day 1 of 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TSST Women Oxytocin | TSST Women Placebo | TSST Men Oxytocin | TSST Men Placebo
Number analyzed (Participants) | 24 | 25 | 32 | 31
units on a scale | 3.08 (3.69) | 3.24 (3.38) | 3.45 (3.35) | 3.45 (3.35)

5. Secondary Outcome: Subject Cocaine Craving MRI 1
Description: as for outcome 4
Time Frame: Subjects rated craving immediately following the first of two MRI scans on Day 2 of 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MRI 1 Women Oxytocin | MRI 1 Women Placebo | MRI 1 Men Oxytocin | MRI 1 Men Placebo
Number analyzed (Participants) | 19 | 23 | 28 | 29
units on a scale | 2.89 (3.31) | 2.65 (2.81) | 3.04 (2.70) | 3.69 (2.99)

6. Secondary Outcome: Subject Cocaine Craving MRI 2
Description: as for outcome 4
Time Frame: Subjects rated craving immediately following the second of two MRI scans on Day 3 of 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MRI 2 Women Oxytocin | MRI 2 Women Placebo | MRI 2 Men Oxytocin | MRI 2 Men Placebo
Number analyzed (Participants) | 23 | 18 | 27 | 28
units on a scale | 2.17 (2.70) | 2.61 (2.78) | 2.04 (2.38) | 2.29 (2.54)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from consent to the 1 month follow-up. That time period ranged from 6 weeks to 3 months.
Arm/Group | TSST Women Oxytocin | TSST Women Placebo | MRI 1 Women Oxytocin | MRI 1 Women Placebo | MRI 2 Women Oxytocin | MRI 2 Women Placebo | TSST Men Oxytocin | TSST Men Placebo | MRI I Men Oxytocin | MRI I Men Placebo | MRI 2 Men Oxytocin | MRI 2 Men Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25 | 0/19 | 0/23 | 0/23 | 0/18 | 0/32 | 0/31 | 0/28 | 0/29 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/19 | 0/23 | 0/23 | 0/18 | 0/32 | 0/31 | 0/28 | 0/29 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/19 | 0/23 | 0/23 | 0/18 | 0/32 | 0/31 | 0/28 | 0/29 | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT01573273/Prot_SAP_000.pdf